CLINICAL TRIAL: NCT00109239
Title: A Multicenter, Open-Label, Phase III, Randomized, Active-Controlled Trial Evaluating the Efficacy, Safety, and Pharmacokinetics of rhuMAb VEGF (Bevacizumab), in Combination With Capecitabine Chemotherapy, in Subjects With Previously Treated Metastatic Breast Cancer
Brief Title: A Study of rhuMAb VEGF (Bevacizumab) in Combination With Chemotherapy in Patients With Previously Treated Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: AVF2119g; NCT00012285 (obsolete NCT alias)
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Metastatic; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Drug: rhuMAb VEGF (Bevacizumab)

SUMMARY:
This Phase III, multicenter, randomized, active-controlled, open-label trial is designed to evaluate the efficacy, safety, and pharmacokinetics of rhuMAb VEGF when combined with capecitabine compared with capecitabine alone in subjects with previously treated metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Women >=18 years of age
* Histologically confirmed carcinoma of the breast with metastatic disease that is currently progressing; in subjects who present with metastatic disease, cytologic confirmation is permissible
* Prior administration of one or two conventional chemotherapy regimens for metastatic disease (Subjects who have had bone marrow or peripheral blood stem cell transplantation in association with chemotherapy are eligible for this study.) -OR-
* No prior chemotherapy for metastatic disease if the subject received a regimen containing both an anthracycline (or anthracenedione) and a taxane as adjuvant therapy and if relapse occurred within 12 months of completing adjuvant chemotherapy
* Prior administration of both an anthracycline (or anthracenedione) and a taxane in either the adjuvant or metastatic setting
* Recovery from reversible toxicities of prior therapy
* Bi-dimensionally measurable disease; at least one target lesion must be bi-dimensionally measurable and at least one target lesion must not have been biopsied recently; all target lesions must be >=2 cm in longest dimension
* ECOG performance status of 0 or 1
* Use of an effective means of contraception in women of childbearing potential
* Life expectancy of >=3 months
* Willingness and capability to be accessible for follow-up

Exclusion Criteria:

* Pleural effusions or bone lesions as the only manifestations of the current metastatic breast cancer
* Known HER2-positive status (either 3+ by immunohistochemistry or positive by FISH), as evaluated at the institution, unless the subject has previously relapsed following Herceptin(R) therapy. Subjects may not continue Herceptin therapy while enrolled in this trial.
* Other primary malignancies (other than basal cell carcinoma of the skin or in situ cervical cancer) within the 5 years preceding Day 0
* Prior radiotherapy to a measurable metastatic lesion(s) if it is to be used as the only lesion to measure response, unless the target lesion within the radiation field is actively progressing and radiotherapy was completed >=6 months prior to randomization
* Radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for metastatic breast cancer within 21 days prior to Day 0
* Use of bisphosphonates unless initiated at least 21 days before Day 0
* Previous treatment with capecitabine
* Previous treatment with rhuMAb VEGF
* History or evidence upon physical examination of CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke; all subjects must have a baseline CT or MRI of the head.)
* Serious, non-healing wound, ulcer, or bone fracture
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year prior to Day 0
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations other than in the breast within 7 days prior to Day 0; placement of a vascular access device within 7 days prior to Day 0

  * Current or recent (within 10 days prior to Day 0) use of full-dose oral or parenteral anticoagulants or thrombolytic agents (except as required to maintain patency of preexisting, permanent indwelling IV catheters; for subjects receiving warfarin, international normalized ratio [INR] of <1.5; appropriate use of heparin should be discussed with the Medical Monitor)
  * Chronic, daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory medications (of the kind known to inhibit platelet function at doses used to treat chronic inflammatory diseases)
* Presence of bleeding diathesis or coagulopathy
* Active infection requiring parenteral antibiotics on Day 0
* Pregnancy (positive pregnancy test) or lactation

  * Proteinuria at baseline or clinically significant impairment of renal function
* Severe renal impairment (creatinine clearance <30 mL/min at baseline using the Cockcroft-Gault formula)
* Known sensitivity to 5-FU
* Lack of physical integrity of the upper gastrointestinal tract, known malabsorption or other significant disease of the stomach, small intestine, liver, or kidney that may adversely affect the pharmacokinetics of capecitabine
* History of allergy to iodine-containing contrast that required treatment and that would prohibit use of CT scan with contrast
* Screening clinical laboratory values: *ANC of <1500/uL; *Platelet count of <75,000/uL; *INR of >=1.5; *Total bilirubin of >1.5 times upper limit of normal; *AST or ALT >2.5 times the upper limit of normal (>5 times the upper limit of normal in subjects with known metastatic disease in the liver); *Serum creatinine of >2.0 mg/dL; *Hemoglobin of <9 gm/dL (may be transfused to maintain or exceed this level)
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Current or recent (within 28 days prior to Day 0) participation in another experimental drug study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Study Completion 2002-09 (Actual)

REFERENCES:
- [Derived] Scappaticci FA, Skillings JR, Holden SN, Gerber HP, Miller K, Kabbinavar F, Bergsland E, Ngai J, Holmgren E, Wang J, Hurwitz H. Arterial thromboembolic events in patients with metastatic carcinoma treated with chemotherapy and bevacizumab. J Natl Cancer Inst. 2007 Aug 15;99(16):1232-9. doi: 10.1093/jnci/djm086. Epub 2007 Aug 8. PMID 17686822